CLINICAL TRIAL: NCT05548348
Title: A Single Arm, Multicenter Study of First-line Furmonertinib Treatment in Patients With Advanced Epidermal Growth Factor Receptor Uncommon Mutation Positive Non-small Cell Lung Cancer
Brief Title: First-line Furmonertinib in Advanced NSCLC Patients With EGFR Uncommon Mutation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chongqing University Cancer Hospital (Other)
Collaborators: Army Specialty Medical Center (Unknown); The Second Affilicated Hospital of Chongqing Medical University (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ChongqingCancer
Record Dates: First submitted 2022-09-13; First posted 2022-09-21 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Non-small Cell Lung Cancer; EGFR G719X; EGFR L861Q; EGFR S768I
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — aflutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Furmonertinib treatment (Experimental): Furmonertinib will be administered orally at a dose of 160 mg per time, Q.D.
  Interventions: Drug: Furmonertinib 160 mg, Q.D.

INTERVENTIONS:
Drug: Furmonertinib 160 mg, Q.D. — Furmonertinib will be administered orally at a dose of 160 mg per time, Q.D.
  Other Names: AST2818 160 mg, Q.D.

SUMMARY:
Furmonertinib, a newly-designed pan-EGFR-TKI with a trifluoroethoxypyridine-based molecule structure, has shown promising clinical efficacy in EGFR Ex19del/L858R/T790M/Ex20ins mutant advanced NSCLC with an acceptable safety profile without new signals from 80mg to 240mg dose level in phase 1-3 clinical trials. Whether EGFR G719X/S768I/L861Q mutation positive advanced NSCLC patients can benefit from first-line furmonertinib 160mg per day has not been reported. This study aims to investigate the efficacy and safety of furmonertinib 160mg per day in EGFR G719X/S768I/L861Q mutant patients under first-line treatment of advanced NSCLC setting.

DETAILED DESCRIPTION:
This is a single arm, multicenter study which will recruit about 30 patients in China.

The study is designed to evaluate the efficacy and safety of furmonertinib in the first-line treatment of patients with EGFR G719X/S768I/L861Q mutations in advanced NSCLC.

Furmonertinib will be administered orally at a dose of 160 mg per time, Q.D.

ELIGIBILITY:
Inclusion Criteria:

* Provide informed consent prior to any study specific procedures;
* 18 -70 years of age;
* ECOG PS of 0 to 1 at screening with no clinically significant deterioration in the previous 2 weeks, life expectancy ≥12 weeks;
* Pathologically confirmed Non-Small Cell Lung Cancer (NSCLC);
* Locally advanced or metastatic NSCLC not amenable to curative surgery or radiotherapy (stage IIIB-IV, according to the 8th edition of the AJCC staging system);
* Patient with EGFR G719X or S768I or L861Q mutation diagnosed histologically or cytologically, the reports must be issued or recognized by Tier 3A hospitals. The mutations above may exist alone or together;
* No previous systemic anti-tumor therapy for locally advanced or metastatic NSCLC;
* According to RECIST 1.1, patients have at least one tumor lesion at baseline that meets the following requirements: accurately and repeatably measurable at baseline have no radiotherapy or biopsy;
* For premenopausal women with childbearing potential, a pregnancy test must be performed within 14 days before the first dose, and the pregnancy test (blood or urine test) must be negative; female subjects must not be lactating;
* Willing to use contraception (male patients); Voluntary and agree to follow the study treatment protocol as well as follow-up plan, and can accept the oral medicine treatment.

Exclusion Criteria:

* small cell lung carcinoma;
* History of hypersensitivity to active or inactive excipients of investigational product (IP) or drugs with a similar chemical structure or class to investigational product (IP);
* Confirmed EGFR Ex20ins or Ex19del or L858R or T790M mutant;
* Patient who receive prior treatment including: any Epidermal growth factor receptor tyrosine kinase inhibitors (EGFR-TKI); the patients who have received intrapleural perfusion therapy can only be enrolled 28 days or more after the pleural effusion is stable; major surgery within 4 weeks of the first dose of investigational product (IP); radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation within 4 weeks of the first dose of IP; CYP3A4 strong inhibitor or strong inducer is used within 7 days prior to the first dose, or need to receive these drugs during the study period; traditional Chinese medicine and traditional Chinese medicine preparations with anti-tumor as indications and with adjuvant treatment of tumor is used within 7 days prior to the first dose, or need to receive these drugs during the study period; patients who are receiving drugs known to prolong QTc interval or may cause torsade de pointe and need to continue to receive these drugs during the study period; the time from the treatment with any other investigational product or its analogue to the first dose does not exceed 5 half-lives of the drug or 14 days, whichever is longer.
* Prior treatment with any systemic anti-cancer therapy for advanced Non-Small Cell Lung Cancer (NSCLC) including chemotherapy, biologic therapy, target therapy, immunotherapy, or any investigational drug, except neoadjuvant or adjuvant therapy before 6 months prior to the first dose IP;
* At the beginning of study treatment, any unresolved toxic reaction to prior treatment is present, which exceeds Grade 1 in accordance with Common Terminology Criteria for Adverse Events (CTCAE) (except for alopecia), and exceeds Grade 2 for prior platinum treatment-related neuropathy;
* Spinal cord compression; symptomatic and unstable brain metastases, except for those patients who have completed definitive therapy, are not on steroids, and have a stable neurological status for at least 2 weeks after completion of the definitive therapy and steroids.
* Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product, or previous significant bowel resection that would preclude adequate absorption of IP;
* Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension, active bleeding diatheses, and active infection, which in the Investigator's opinion makes it undesirable for the patient to participate in the trial;
* Past medical history of Interstitial Lung Disease (ILD), drug-induced Interstitial Lung Disease, radiation pneumonitis that required steroid treatment, or any evidence of clinically active Interstitial Lung Disease;
* Any evidence of corneal injury;
* Inadequate bone marrow reserve or organ function;
* QT prolongation or any clinically important abnormalities in rhythm and heart function;
* Pregnancy or lactation;
* Patients who may have poor compliance with the research procedures and requirements, etc., as judged by investigators.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-09-26 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Approximately 12 months from the first patient begin study treatment
  Objective Response Rate (ORR) (per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) using Investigator assessments) is defined as the number (%) of patients with response of Complete Response or Partial Response. Data obtained up until progression, or the last evaluable assessment in the absence of progression, will be included in the assessment of Objective Response Rate.

SECONDARY OUTCOMES:
Disease Control Rate (DCR) by Investigator | Approximately 12 months from the first patient begin study treatment
  Disease control rate (DCR) is defined as the percentage of subjects who have a best overall response of Complete Response (CR) or Partial Response (PR) or Stable Disease (SD) by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) as assessed by the Investigator.
Progression-free survival (PFS) | Approximately 24 months after the first patient begin study treatment.
  Progression-free survival (PFS) using Investigator assessment as defined by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1). Progression-free survival (PFS) is defined as the time from beginning of study treatment until the date of objective disease progression or death (by any cause in the absence of progression). Patients who have not progressed or died at the time of analysis will be censored at the time of the latest date of assessment from their last evaluable Response Evaluation Criteria in Solid Tumors (RECIST) assessment.
Duration of Response (DoR) | Duration of Response analysis will occur when Progression-free survival (PFS) maturity is observed at approximately 24 months from the first patient begin study treatment
  Duration of Response is defined as the time from the date of first documented response until the date of documented progression or death in the absence of disease progression.
Overall Survival (OS) | The analysis of OS will be conducted at 2 time points: when PFS maturity is observed at approximately 24 months after the first patient begin study treatment, and when OS maturity is observed at approximately 36 months after the first patient begin study
  Overall survival is defined as the time from beginning of study treatment until death due to any cause.
Adverse Events | From the start of study drug to 30 days after the last dose of study drug
  The number of patients with adverse events and the severity according to CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Yongsheng Li, M.D. & Ph.D., Principal Investigator — Chongqing University Cancer Hospital
Locations (3):
- China (3):
  - The Second Affilicated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - Army Specialty Medical Center, Chongqing, Chongqing Municipality

IPD SHARING:
Plan to Share IPD: No